CLINICAL TRIAL: NCT06836817
Title: Voice and Behcet's Disease
Brief Title: Evaluation of Voice in Behcet's
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Wafaa Helmy Abdelhakeem, doctor, Minia University
Other Study IDs: voice in Behcet's Disease
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Behcet Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I: Group I will comprise of the 30 patients with Behçet's disease (BD).
  Interventions: Other: 1-Laryngyscopic examination 2-Acoustic analysis
- Group II: Group II will comprise of 30 controls.
  Interventions: Other: 1-Laryngyscopic examination 2-Acoustic analysis

INTERVENTIONS:
Other: 1-Laryngyscopic examination 2-Acoustic analysis — 1. History taking.
  2. voice sample by recording (in sustained vowel |a| )
  3. Auditory Perceptual Assessment (APA): (Kotby et al., 1986)
  4. Laryngyscopic examination:
     Patients will taken to a room with a tower on which the 8.5 mm 70 rigid laryngoscope (KARL STORZ - endoscope) (Tele pack X LED).
  5. Acoustic analysis: The voice sample will be subjected to computerized acoustic analysis using Multidimensional voice program software(MDVP).

SUMMARY:
Behçet's disease (BD) is a systemic inflammatory condition of unknown origin with no definite aetiopathogenetic pathways accepted worldwide. To date, only a few studies have investigated laryngeal involvement in BD and data about this are scarce. For these reasons, the present study focuses on verifying the occurrence of vocal cord involvement in patients with BD, identifying potential correlations with specific demographic, clinical, and therapeutic characteristics.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a systemic inflammatory condition of unknown origin with no definite aetiopathogenetic pathways accepted worldwide. BD owes its name to the Turkish dermatologist Hulusi Behçet, whom published in 1937 two cases of oral aphthous, genital ulcers, and recurrent uveitis with hypopion, known as triple-symptom complex. In addition to these, other clinical features encompass musculoskeletal, gastrointestinal, renal, pulmonary, cardiovascular, and cutaneous manifestations including erythema nodosum and pseudofolliculitis.To date, only a few studies have investigated laryngeal involvement in BD and data about this are scarce. For these reasons, the present study focuses on verifying the occurrence of vocal cord involvement in patients with BD, identifying potential correlations with specific demographic, clinical, and therapeutic characteristics.The study will include 60 volunteers. They will divided into 2 groups. Group I will comprise of the 30 patients with Behçet's disease (BD), and Group II will comprise of 30 controls.The inclusion criteria for selection of Group I participants will based on the criteria of the International Study Group which was proposed in 1990. The inclusion criteria for Group II will not have a Behcet's Disease.Methods

1. History taking.
2. voice sample by recording (in sustained vowel |a| )
3. Auditory Perceptual Assessment (APA): (Kotby et al., 1986)
4. Laryngyscopic examination:

   Patients will taken to a room with a tower on which the 8.5 mm 70 rigid laryngoscope (KARL STORZ - endoscope) (Tele pack X LED).
5. Acoustic analysis: The voice sample will be subjected to computerized acoustic analysis using Multidimensional voice program software(MDVP).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for selection of Group I participants will based on the criteria of the International Study Group which was proposed in 1990. The inclusion criteria for Group II will not have a Behcet's Disease.

Exclusion Criteria:

* other autoimmune diseases.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 60 volunteers. They will divided into 2 groups. Group I will comprise of the 30 patients with Behçet's disease (BD), and Group II will comprise of 30 controls.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
laryngoscopic pictures | baseline
  abnormal anatomical laryngeal findings like laryngeal congestion, bleeding, vocal fold polyps, cysts, nodules
frequency | baseline
  frequency in hertz
jitter | baseline
  jitter in percentage %
shimmer | baseline
  shimmer in decibl
harmonic to noise ratio | baseline
  harmonic to noise ratio in decibl

IPD SHARING:
Plan to Share IPD: Undecided